CLINICAL TRIAL: NCT01746550
Title: A Single Arm Clinical Trial in Japan for Reconstruction of Obstructive Lesions of the Superficial Femoral Artery or Proximal Popliteal Artery by Bard LifeStent.
Brief Title: A Safety and Effectiveness Study of the MD-12-001 Stent in the Treatment of Superficial Femoral Artery or Popliteal Artery Blockages in Japanese Patients
Acronym: Reliable
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Collaborators: Medicon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MED-12-001
Record Dates: First submitted 2012-12-07; First posted 2012-12-11 (Estimated); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Arterial Occlusive Disease
MeSH Terms: conditions — Arterial Occlusive Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MD-12-001 Stent Arm (Experimental): This study includes a single arm, the MD-12-001 Stent Arm.
  Interventions: Device: MD-12-001 Stent

INTERVENTIONS:
Device: MD-12-001 Stent — MD-12-001 is a self-expanding nitinol stent
  Other Names: Bard Lifestent Vascular Stent

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of the MD-12-001 stent in the treatment of superficial femoral artery and proximal popliteal artery blockages in Japanese patients.

ELIGIBILITY:
Key Inclusion Criteria:

* Rutherford Category 2-4 (mild intermittent claudication (pain while walking)to ischemic pain (pain due to decreased blood flow) at rest).
* The target lesion(s) has evidence of narrowing or blockage and can be stented.
* The total length of the lesion or series of lesions is estimated to be less than or equal to 150 mm.
* The target vessel reference diameter is greater than or equal to 4.0 mm and less than or equal to 6.5 mm

Key Exclusion Criteria:

* The subject has a known reaction (including allergic reaction) or sensitivity to blood thinning medications, or study device materials (nickel, titanium or tantalum)
* The subject has a known sensitivity to medical imaging substances (contract media) that cannot be pretreated with medications (steroids or/and antihistamines)
* The subject has a history of bleeding disorders (diatheses or coagulopathy).
* The subject has kidney failure or is having dialysis treatment.
* The subject has insufficient liver function, swelling of vein(s) caused by blood clot (thrombophlebitis), uremia, systemic lupus, or deep vein blood clots.
* Subject has Acute Limb Ischemia (a sudden loss of blood flow to the limb).
* Subject has a history of bypass surgery on the study vessel.
* Subject has a history of heart attack or stroke within 6 months of study procedure.
* The subject is receiving immunosuppressive therapy (medications that lower the body's normal immune response).
* The subject is diagnosed with a severe infection (septicemia).
* Principal investigator determines the subject's condition would prevent the subject from undergoing the study procedure or cannot support a vascular bypass graft.
* The subject with a stent previously implanted into the target vessel.
* Subject has disease in both legs where both limbs meet the inclusion criteria and it is planned to treat both limbs within 30 days.
* Pregnant, possibly pregnant and/or nursing female subjects are excluded, as are female subjects who are willing to have a baby during the trial.
* The subject is participating in an investigational drug or another investigational device study.
* Subject has a large amount of blood clot next to the study lesion.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-12; Primary Completion 2014-10-11 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects who are free of target limb failure at 12-months post study procedure. | 12-months post study procedure

SECONDARY OUTCOMES:
The proportion of subjects who are free of target limb failure. | 30-days, 6-, 24-, and 36-months post study procedure
The proportion of subjects with primary target lesion patency. | 30-days, 6-, 12-, 24-, and 36-months post study procedure
  This endpoint will assess whether the study blockage has been unblocked using ultrasound imaging assessments reviewed by an independent core laboratory.
The proportion of subjects with secondary target vessel/lesion patency. | 30-days, 6-, 12-, 24-, and 36-months post study procedure
  This endpoint will assess whether the study blockage has shut again; where the target vessel/lesion no longer has blood flow or where surgical bypass of the vessel is performed.
Proportion of subjects who achieve acute procedural success. | Perioperative period (period during study procedure)
Rutherford category assessment. | Baseline, 30-days. 3-. 6-. 12-. 24-. 36-. 48- and 60-months post study procedure
  The assessment of peripheral artery disease severity will be performed using the Rutherford Classification system.
Ankle-brachial index measurements. | Baseline, 30-days, 3-, 6-, 12-, 24-, 36-, 48-, and 60-months post study procedure
  The ratio of blood pressure in the lower legs to the blood pressure in the arms will be calculated and assessed as a measure of disease severity.
Quality of Life (SF-36) Questionnaire | Baseline, 30-days, 3- , 6-, 12-, 24-, 36-, 48-, and 60-months post study procedure
  The SF-36 Quality of Life Questionnaire (QOL) will be used to evaluate QOL changes during study participation.
Proportion of Subjects who experience Major Adverse Events. | 30-days post procedure
  Major Adverse Events is defined as any death, stroke, myocardial infarction (heart attack) or target limb amputation.
Proportions of Subjects who experience 1) any adverse event and 2) any serious adverse event. | through 60-months post study procedure
The proportion of subjects who undergo target vessel/lesion revascularization (restoration of blood flow) | 12-, 24-, 36-, 48-, and 60-months post study procedure
Proportion of subjects without stent fracture | 30-days, 6-, 12-, 24, and 36-months post study procedure

CONTACTS AND LOCATIONS:
Overall Officials: Masato Nakamura, Principal Investigator — Toho University Ohashi Hospital
Locations (12):
- Japan (12):
  - Kokura Kinen, Kitakyushu, Fukuoka
  - Tokeidai Hospital, Sapporo, Hokkaido
  - Kansai Rosai Hospital, Amagasaki, Hyōgo
  - Shonankamakura General Hospital, Kamakura, Kanagawa
  - Saiseikai Yokohamashi Tobu Hospital, Yokohama, Kanagawa
  - Sendai Kousei Hospital, Sendai, Miyagi
  - Nara Medical University Hospital, Kashihara, Nara
  - Kishiwada Tokushukai Hospital, Kishiwada, Osaka
  - Kasukabe Chuo General Hospital, Kasukabe, Saitama
  - Toho University Ohashi Hospital, Meguro City, Tokyo
  - The Jikei University Hospital, Minato, Tokyo
  - Kyushu University Hospital, Fukuoka